CLINICAL TRIAL: NCT05435742
Title: A Randomized, Double-blind, Placebo-controlled Phase 1b/2a Study to Evaluate the Safety, Tolerability, and Efficacy of Repeated Subcutaneous Administration of SON-080 in Patients With Persistent Chemotherapy-induced Peripheral Neuropathy (CIPN) After the End of Chemotherapeutic Treatment
Brief Title: SON-080 in Patients With Persistent Chemotherapy-induced Peripheral Neuropathy (CIPN)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Sonnet BioTherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB211
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SON-080 Dose Level 1 (Experimental): 20 µg SON-080 SC administration TIW
  Interventions: Biological: SON-080
- SON-080 Dose Level 2 (Experimental): 60 µg SON-080 SC administration TIW
  Interventions: Biological: SON-080
- Matching Placebo (Placebo Comparator): Matching placebo 20 µg SON-080 SC administration TIW
  Interventions: Biological: SON-080

INTERVENTIONS:
Biological: SON-080 — Recombinant human interleukin-6 (rhIL-6)

SUMMARY:
The study will be conducted in adult patients with Chemotherapy-induced Peripheral Neuropathy (CIPN) that has been persistent for at least 3 months following completion of chemotherapy. A total of 60 patients will be enrolled in equal numbers of a placebo group and two different SON-080 dose groups. Treatment period will be 12 weeks long and patients will be followed-up for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, inclusive, at the time of Screening.
* Have persistent CIPN at 3 months or more after chemotherapeutic treatment arrest (QLQ-CIPN20 score of 30 to 100).
* Have a history of cancer that is stable or in remission at the time of study entry.
* Have a history of treatment with a chemotherapeutic agent in the taxane, organoplatin, or vinca alkaloid family.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 at Screening.
* Must have adequate organ function, defined as:

  * Hematologic function defined as National Cancer Institute (NCI) CTCAE Grade 1 or less for all blood parameters.
  * Renal function defined as calculated creatinine clearance or radioisotope glomerular filtration rate >60 mL/min/1.73 m2 or normal serum creatinine with a maximum serum creatinine of 1.7 mg/dL for males and 1.4 mg/dL for females.
  * Hepatic Function defined as:
  * Alanine aminotransferase (ALT) ≤3 × the upper limit of normal (ULN) for age.
  * Total bilirubin ≤1.5 × ULN (unless the patient has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin).
* Either the patient or the caregiver must be willing and able to administer SC treatment in an at-home setting after training.
* Female patients of childbearing potential who are not currently pregnant or lactating must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β HCG]) on day 1 and agree to abstinence or use a highly effective method of birth control for 30 days before the study, during the study, and for 30 days after the last dose of study intervention. Females who are not of childbearing potential (have had a tubal ligation, hysterectomy, or bilateral oophorectomy, or are ≥ 1-year postmenopause) or have a partner who has had a vasectomy do not need to use any contraception.
* Nonchildbearing potential is defined as surgically sterile (documented hysterectomy, tubal ligation, or bilateral salpingo-oophorectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea). If necessary, a follicle-stimulating hormone (FSH) level ≥ 35 IU/L at Screening will be considered confirmatory in the absence of a clear postmenopausal history. If a patient is not sexually active, but becomes active, then she and her male partner must use adequate contraception.
* Male patients and their female partners must agree to use adequate contraception (including a barrier method) during the study and for 30 days after the last dose of SON-080. Contraception guidance is described in the protocol.
* If a patient is not sexually active, but becomes active, then he and his female partner must use adequate contraception. Male patients must refrain from sperm donation for 90 days after the last dose of SON-080.
* Must be willing and able to provide voluntary written informed consent to participate in the study.
* Must be able to communicate well with the Investigator and/or study site personnel and to comply with the requirements of the entire study.

Exclusion Criteria:

* Evidence of current alcohol or drug dependence.
* Evidence for other cause of chemotherapeutic neuropathy, e.g., use of colchicine, amiodarone, thalidomide, vitamin B12 deficiency, etc.
* Unresolved toxicities from prior anticancer therapy, defined as not having resolved to baseline or to CTCAE Grade 1, except for alopecia, or to the levels dictated in the inclusion/exclusion criteria.
* Active infection with SARS-CoV-2, as determined by local SOPs for testing during Screening.
* History of hepatic disease or active clinically significant liver function test results, defined as chronically abnormal ALT, aspartate aminotransferase (AST), total bilirubin and fractionated bilirubin, and alkaline phosphatase >1.5 × the ULN. Note: Isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%.
* Diagnosis of or positive screening result for hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV)-1 or HIV-2.
* Known allergies to any of the ingredients of the medicinal product or to acetaminophen.
* History of brain metastases.
* Diagnosed with lymphoma, Kaposi's sarcoma, or multiple myeloma.
* Significant unstable vascular disease, as judged by the Investigator.
* Any other investigational drug in the 4 weeks preceding treatment administration. Note: COVID-19 vaccines will be allowed if administered more than 14 days before the first dose administration.
* Clinical history of a thrombosis, deep vein thrombosis, or pulmonary embolus in the past year.
* Other serious concurrent medical condition which, in the opinion of the Investigator, would preclude inclusion in the study.
* History of any active infection within 14 days before the first dose of SON-080, if deemed clinically significant by the Investigator and Sponsor.
* Concurrent conditions that could interfere with safety and/or tolerability measurements.
* Pregnant and/or lactating.
* Unable or unwilling to cooperate with the Investigator for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of SON-080 | Through study completion, an average of 24 weeks
  Frequency and severity of treatment emergent adverse events (TEAEs), including serious adverse events (SAEs) and deaths, by treatment. Note that progression of, or death from, the underlying tumor will not be considered an SAE.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of SON-080 | Through study completion, an average of 24 weeks
  Single- and multiple-dose PK parameters of SON-080
Evaluate the immunogenicity of SON-080 | Through study completion, an average of 24 weeks
  Anti-SON-080 antibody determination
Evaluate the preliminary efficacy of SON-080 | Weeks 5, 9, and 12 of treatment, as well as 4 and 12 weeks after the end of treatment.
  Change from baseline in Quality-of-Life Questionnaire-CIPN 20-item scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kenney, MD, Study Director — Sonnet BioTherapeutics
Locations (1):
- Emeritis Research, Camberwell, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Baat A, Trinh B, Ellingsgaard H, Donath MY. Physiological role of cytokines in the regulation of mammalian metabolism. Trends Immunol. 2023 Aug;44(8):613-627. doi: 10.1016/j.it.2023.06.002. Epub 2023 Jul 7. PMID 37423882